CLINICAL TRIAL: NCT03090074
Title: To Lower Glucose Levels and Reduce Weight by Exclusion of Carbohydrates and Inclusion of Psychological Behavioral Support
Brief Title: Moderate or Extensive Carbohydrate Reduction in Risk Patients
Acronym: LOWinCHIP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Fredrik H Nystrom, Professor, head of Internal Medicine, consultant in Endocrinology., University Hospital, Linkoeping
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LOWinCHIP
Record Dates: First submitted 2017-03-20; First posted 2017-03-24 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Glucose Metabolism Disorders
MeSH Terms: conditions — Glucose Metabolism Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Moderate carbohydrate restriction and traditional support (Active Comparator): Moderate carbohydrate restriction and traditional support with group meetings
  Interventions: Behavioral: Diet regime; Behavioral: Type of psychological support
- Extreme low carbohydrate diet and traditional support (Active Comparator): Extreme carbohydrate restriction and traditional support with group meetings
  Interventions: Behavioral: Diet regime; Behavioral: Type of psychological support
- Moderate carbohydrate restriction and ACT support (Active Comparator): Moderate carbohydrate restriction and psychological support based on acceptance and commitment therapy
  Interventions: Behavioral: Diet regime; Behavioral: Type of psychological support
- Extreme carbohydrate restriction and ACT support (Active Comparator): Extreme carbohydrate restriction and psychological support based on acceptance and commitment therapy
  Interventions: Behavioral: Diet regime; Behavioral: Type of psychological support

INTERVENTIONS:
Behavioral: Diet regime — Randomization to moderate or extreme low-carbohydrate Mediterranean diet advice.
Behavioral: Type of psychological support — Randomization to group-based psychological support according to ACT or to traditional cognitive behavioral therapy

SUMMARY:
Risk-patients for diabetes or patients that are diagnosed with this condition but who are not treated with insulin are randomized two times, according to diet and according to the type of support:

Randomization with regard to carbohydrate restriction (25-30 E% or < 10E%). Randomization with regard to type of psychological support. Either according to Acceptance and Commitment Therapy or to traditional cognitive behavioral therapy. Both kinds of psychological support is given as group therapy.

Two-hundred patients are recruited and each patient is followed for two years.

DETAILED DESCRIPTION:
The organizers will recruit 200 patients in the study "To lower glucose levels and reduce weight by exclusion of carbohydrates and inclusion of psychological behavioral support" (LOWinCHIP) at the primary care health center "Cithyhälsan Centrum" in Norrköping. Each patient will be followed for 2 years. Patients are eligible if they have are above 18 years of age and have a BMI above 28 kg/m2 and also belong to one or more of the following groups: 1) type 2 diabetes that is not treated with insulin. 2) Patients that have had gestational diabetes or who have 3) first grade relative with type 2 diabetes. Finally 4) pre-diabetic individuals with impaired fasting glucose (6.1-6.9 mmol) or impaired glucose tolerance (capillary plasma glucose 8.9-12-1 after glucose challenge) are also potential participants. Patients must not have insulin therapy or severe kidney failure (GFR< 30). They can also not have severe physical restrictions for activity and they must not have difficulties with understanding written Swedish texts.

The participants are randomized two times (two by two factorial):

Randomization with regard to carbohydrate restriction (25-30 E% or < 10E%). Randomization with regard to type of psychological support. Either according to Acceptance and Commitment Therapy (ACT) or to traditional cognitive behavioral therapy. Each group will have three group sessions with approximately 8 participants followed by a telephone call by the therapist. Each session will be held by the psychologists that are part of the Cityhälsan Centrum staff.

The study has > 95% power to demonstrate 5% HbA1c (mmol/mol) difference between groups with a drop out of 25%.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes without insulin. Patients at high risk for developing diabetes.

Exclusion Criteria:

* Severe kidney failure. Insulin therapy. Inability to understand instructions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-03-20 (Actual); Primary Completion 2021-03-19 (Estimated); Study Completion 2021-03-19 (Estimated)

PRIMARY OUTCOMES:
Long-term glucose levels | 2 years
  HbA1c levels

SECONDARY OUTCOMES:
Quality of Life | 2 years
  Quality of Life by questionnaires
Cardiovascular risk factors | 2 years
  Lipids, body weight, glucose, ketones

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Linkoping, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: No
It is not planned to be shared